CLINICAL TRIAL: NCT01449396
Title: Chinese Traditional Medicine Contribution to Improve In-vitro Fertilization (IVF) Results: Acupuncture in Embryo Transfer
Brief Title: Acupuncture, Chinese Traditional Medicine, in Embryo Transfer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACU2010
Record Dates: First submitted 2011-10-04; First posted 2011-10-10 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Pregnancy
Keywords: acupuncture; in vitro fertilization; embryo transfer
MeSH Terms: interventions — Bed Rest; Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- SHAM ACUPUNCTURE (Sham Comparator): Sham intervention: acupuncture needle without puncture nor stimulation
  Interventions: Procedure: Acupuncture
- REAL ACUPUNCTURE (Experimental): Experimental: acupuncture in selected points of the protocol designed
  Interventions: Procedure: Acupuncture
- Control (Other): Bed Rest
  Interventions: Other: Bed Rest

INTERVENTIONS:
Other: Bed Rest — Bed rest during 25 minutes on day 1, 4 and 6 of ovarian stimulation, before and after embryo transfer
  Arms: Control
Procedure: Acupuncture — Sham acupuncture during 25 minutes on day 1, 4 and 6 of ovarian stimulation, before and after embryo transfer
  Arms: SHAM ACUPUNCTURE
Procedure: Acupuncture — Acupuncture during 25 minutes on day 1, 4 and 6 of ovarian stimulation, before and after embryo transfer
  Arms: REAL ACUPUNCTURE

SUMMARY:
The aim of the study is to prove that acupuncture applied before and after embryo transfer is able to increase pregnancy rates by means of reducing stress and improving endometrial vascularization in women receiving in vitro Fertilization (IVF) treatments.

DETAILED DESCRIPTION:
Around 75% of all in vitro fertilization (IVF) treatments fail in providing a healthy baby at home. Most of the women undergoing those techniques suffer in some extent anxiety, depression and stress. Stress make IVF results worse and it has been prove by correlating cortisol, adrenaline and noradrenaline levels with failed cycles. Acupuncture has proved its ability to reduce stress levels. Moreover, Acupuncture has prove to have an effect inhibitory on the sympathetic system and this capacity improves vascularization in uterus and ovaries. Available literature concerning these two issues is not conclusive because of studies design. Acupuncture´s biological mechanism on controlled ovarian stimulation and embryo transfer has not been completely described; if it really has one. Published studies show very different designs and inconclusive/contradictory results can be withdrawn making very difficult to take the clinical decision of recommending acupuncture or not to in vitro fertilization (IVF) patients. If acupuncture really enhance pregnancy rates in IVF cycles still unanswered given that no randomized three arms study comparing no intervention to sham acupuncture to acupuncture has been published.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 37 years old
* 18-28 Body mass index (BMI)
* Medical indication of intracytoplasmic sperm injection (ICSI) treatment to treat sterility
* No previous in vitro fertilization (IVF) or intracytoplasmic sperm injection (ICSI) treatments
* No previous experience of acupuncture treatments
* At least one high quality embryo in the day of uterine transfer

Exclusion Criteria:

* Polycystic ovarian syndrome
* Endometriosis
* Reproductive surgeries: any on uterus, fallopian tubes or ovaries
* Ovarian cysts >20mm at the beginning of the stimulation cycle
* Hormone treatment in the previous three months of the stimulation cycle, including oral contraceptives
* Previous miscarriages and ectopic pregnancies
* Coasting
* Oestradiol levels >3500pg/ml or ovarian size >65mm in human chorio gonadotropin (hCG) day.
* Failure to keep confidentiality
* Concomitant illness or severe adverse reaction

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 286 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Pregnancy rate | 14 days after embryo transfer
  Heart beating in intrauterus embryo

SECONDARY OUTCOMES:
Rating preconceived ideas about acupuncture | From 24 hours (h) to 14 days after embryo transfer
  Rating preconceived ideas about acupuncture
Determination of serum prolactin and 24h urine cortisol. | The day of embryo transfer (+14 days post-cycle start)).
  Determination of serum prolactin and 24h urine cortisol to measure stress levels on the day of embryo transfer.
Endometrial vascularization study | The day of embryo transfer (+14 days after cycle start) and 2 days before and after it.
  Endometrial vascularization study on the day of embryo transfer, 2 days before and after it
Analysis of the results of assisted reproductive cycle | After 14 days post-transfer (28 days after cycle star)
  Analysis of the results of assisted reproductive cycle on levels of beta human chorionic gonadotropin (BhCG) +14 days post-transfer, evidence of intrauterine gestational sac with heartbeat and embryo live birth at home

CONTACTS AND LOCATIONS:
Overall Officials: Monica Romeu, Doctor, Principal Investigator
Locations (1):
- Human Reproduction Unit of the University and Politechnic Hospital La Fe., Valencia, Spain

REFERENCES:
- [Background] Dong J. Research on the reduction of anxiety and depression with acupuncture. Am J Acupunct 1993; 21: 327-30.
- [Background] Stener-Victorin E, Waldenstrom U, Andersson SA, Wikland M. Reduction of blood flow impedance in the uterine arteries of infertile women with electro-acupuncture. Hum Reprod. 1996 Jun;11(6):1314-7. doi: 10.1093/oxfordjournals.humrep.a019378. PMID 8671446
- [Background] Paulus WE, Zhang M, Strehler E, El-Danasouri I, Sterzik K. Influence of acupuncture on the pregnancy rate in patients who undergo assisted reproduction therapy. Fertil Steril. 2002 Apr;77(4):721-4. doi: 10.1016/s0015-0282(01)03273-3. PMID 11937123
- [Background] Paulus E, Zhang M Strehler E, Sterzik K. Motility of the endometrium after acupuncture treatment. Fertil Steril 2003; 80 (Suppl 3): 131.
- [Background] Smith C, Coyle M, Norman RJ. Influence of acupuncture stimulation on pregnancy rates for women undergoing embryo transfer. Fertil Steril. 2006 May;85(5):1352-8. doi: 10.1016/j.fertnstert.2005.12.015. Epub 2006 Apr 5. PMID 16600225
- [Background] Dieterle S, Ying G, Hatzmann W, Neuer A. Effect of acupuncture on the outcome of in vitro fertilization and intracytoplasmic sperm injection: a randomized, prospective, controlled clinical study. Fertil Steril. 2006 May;85(5):1347-51. doi: 10.1016/j.fertnstert.2005.09.062. Epub 2006 Apr 17. PMID 16616748
- [Background] Westergaard LG, Mao Q, Krogslund M, Sandrini S, Lenz S, Grinsted J. Acupuncture on the day of embryo transfer significantly improves the reproductive outcome in infertile women: a prospective, randomized trial. Fertil Steril. 2006 May;85(5):1341-6. doi: 10.1016/j.fertnstert.2005.08.070. Epub 2006 Apr 5. PMID 16600232
- [Background] Domar AD, Meshay I, Kelliher J, Alper M, Powers RD. The impact of acupuncture on in vitro fertilization outcome. Fertil Steril. 2009 Mar;91(3):723-6. doi: 10.1016/j.fertnstert.2008.01.018. Epub 2008 Mar 7. PMID 18314118
- [Background] Benson M, ElKind-Hirsch K, Theall A, Fong K, Hogan R, Scott R. Impact of the acupuncture before and after embryo transfer on the outcome of in vitro fertilization cycles: a prospective single blind randomised
- [Background] Craig L, Criniti A, Hansen K, Marshall L, Soules M. Acupuncture lowers pregnancy rates when performed before and after embryo transfer. Fertil Steril 2007; 88 (Suppl 1): S40.
- [Background] Magarelli P, Criddenda D. Acupuncture and IVF poor responders: a cure? Fertil Steril 2004; 81: S20.
- [Background] Magarelli ´P, Cohen M, Criddenda D. Acupuncture and good prognosis IVF patients: synergy. Fertil Steril 2004; 82: S80-1.
- [Background] Magarelli P, Cohen M, Criddenda D. Acupuncture: impact on pregnancy outcomes in IVF patients. 12th World Congress on Human Reproduction, Venice, Italy, March 2005.
- [Background] Magarelli P, Cohen M, Criddenda D. Improvement of IVF outcomes by acupuncture: are egg and embryo qualities involved? Fertil Steril 2005; 83: S9.
- [Background] 15.- Criddenda D, Magarelli P, Cohen M. Acupuncture and in vitro fertilization: does the number of treatments impact reproductive outcomes? Society for Acupuncture Research 2005.
- [Background] Magarelli P, Criddenda D, Cohen M. Proposed mechanism of action of acupuncture on IVF outcomes. Fertil Steril 2006; 86: S174-5.
- [Background] Magarelli P, Criddenda D, Cohen M. The demographics of acupuncture´s impact on IVF outcomes: infertility diagnosis and SART/CDC/age groups. Fdertil Steril 2007; 87: S10-1.
- [Background] El-Toukhy T, Sunkara SK, Khairy M, Dyer R, Khalaf Y, Coomarasamy A. A systematic review and meta-analysis of acupuncture in in vitro fertilisation. BJOG. 2008 Sep;115(10):1203-13. doi: 10.1111/j.1471-0528.2008.01838.x. Epub 2008 Jul 23. PMID 18652588
- [Background] Manheimer E, Zhang G, Udoff L, Haramati A, Langenberg P, Berman BM, Bouter LM. Effects of acupuncture on rates of pregnancy and live birth among women undergoing in vitro fertilisation: systematic review and meta-analysis. BMJ. 2008 Mar 8;336(7643):545-9. doi: 10.1136/bmj.39471.430451.BE. Epub 2008 Feb 7. PMID 18258932
- [Background] Ng EH, So WS, Gao J, Wong YY, Ho PC. The role of acupuncture in the management of subfertility. Fertil Steril. 2008 Jul;90(1):1-13. doi: 10.1016/j.fertnstert.2008.02.094. Epub 2008 Apr 28. PMID 18440533
- [Background] Cheong YC, Hung Yu Ng E, Ledger WL. Acupuncture and assisted conception. Cochrane Database Syst Rev. 2008 Oct 8;(4):CD006920. doi: 10.1002/14651858.CD006920.pub2. PMID 18843737
- [Background] So EW, Ng EH, Wong YY, Lau EY, Yeung WS, Ho PC. A randomized double blind comparison of real and placebo acupuncture in IVF treatment. Hum Reprod. 2009 Feb;24(2):341-8. doi: 10.1093/humrep/den380. Epub 2008 Oct 21. PMID 18940896
- [Background] White AR. A review of controlled trials of acupuncture for women's reproductive health care. J Fam Plann Reprod Health Care. 2003 Oct;29(4):233-6. doi: 10.1783/147118903101197863. PMID 14662058